CLINICAL TRIAL: NCT01408732
Title: Office-sclerotherapy for Epistaxis Due to Hereditary Hemorrhagic Telangiectasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: American Rhinologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1101M95232
Record Dates: First submitted 2011-07-01; First posted 2011-08-03 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Epistaxis; Hereditary Hemorrhagic Telangiectasia
Keywords: Epistaxis; Hereditary Hemorrhagic Telangiectasia; HHT; Sclerotherapy; Epistaxis (nosebleeds) due to Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Epistaxis; Telangiectasia, Hereditary Hemorrhagic | interventions — Sclerotherapy; Sodium Tetradecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment then Sclerotherapy Intervention (Experimental): The standard treatment group will continue their pre-study "standard treatment" methods to treat epistaxis on the first 6 weeks of the study, followed by intervention with sclerotherapy on the second 6 weeks of the study, plus any additionally needed standard treatments for breakthrough epistaxis. Wash out period 2 weeks
  Interventions: Drug: Sclerotherapy; Other: Standard Treatment
- Sclerotherapy Intervention then Standard Treatment' (Experimental): This group will receive, on the first 6 weeks of the study, sclerotherapy with STS to any visible lesions in the nose at the outset, followed by any needed standard treatments for breakthrough epistaxis. On the second 6 weeks of the study this group will continue with standard treatments that they had been receiving for epistaxis prior to the study. Wash out period of two weeks
  Interventions: Drug: Sclerotherapy; Other: Standard Treatment

INTERVENTIONS:
Drug: Sclerotherapy — 3% Sodium tetradecyl sulfate (STS) is mixed with air at a ratio of 4 parts air to 1 part STS for injection into the affected vessels in the nose. Topical anesthetic is applied to the nasal mucosa prior to injections. Once the mixture is ready for injection, the needle is placed into the vessel, in a submucosal fashion, penetrating 1-2 mm, and very small quantities of foam are injected The amount of foam injected into each lesion varies between 0.1 cc to 0.25 cc. Individual injection amounts vary between lesions, patients and treatment sessions. No more than a total of 3 ml of solution is used in each session. During each session, several lesions can be treated, but the total amount of STS used does not exceed 3 cc.
  Other Names: Sotradecol
Other: Standard Treatment — Normal standard of care followed by Drug interevention

SUMMARY:
The purpose of this study is to test a novel and tolerable office-based treatment method, sclerotherapy with sodium tetradecyl sulfate, for recurrent epistaxis (nosebleeds) related to Hereditary Hemorrhagic Telangiectasia (HHT) disease.

DETAILED DESCRIPTION:
Ninety percent of patients who suffer from Hereditary Hemorrhagic Telangiectasia (HHT) experience epistaxis which can range from mild to recurrent, severe, life threatening episodes. Current methods to treat significant epistaxis have limitations, namely the need for general anesthesia and repeated treatments. The objective of this study is to test a novel and tolerable office-based treatment method, sclerotherapy with sodium tetradecyl sulfate (STS), for recurrent epistaxis related to HHT.

Sclerotherapy is the treatment of vascular lesions by injection with an agent which causes thickening of the vessel wall, obstruction of blood flow, clot formation and collapse of the lesion. Sclerotherapy is an established treatment modality for vascular malformations in the skin, GI tract, genitourinary tract and has been used for lesions in various sites in the head and neck. STS is an anion surfactant (detergent) that is commonly used for sclerotherapy. There are case reports in the literature describing sclerotherapy treatments for epistaxis related to HHT using other agents, but these case reports did not lead to prospective studies. We have performed a pilot study to analyze the tolerability and effectiveness of sclerotherapy with STS in a series of patients with recurrent epistaxis related to HHT. In our series, the treatment was found to be well tolerated and effective, based on patient administered questionnaire and review of clinical data. No complications related to the procedure were noted. Further prospective studies would help elucidate the role of sclerotherapy with STS in the treatment algorithm for recurrent epistaxis related to HHT.

Our goal is to conduct a prospective, randomized-controlled trial to test the efficacy and tolerability of sclerotherapy using STS in the treatment of recurrent epistaxis due to HHT. A modified crossover design will be utilized with the intervention group receiving sclerotherapy, plus any additional, previously utilized standard treatment methods needed to control epistaxis. The control group will receive their current standard treatment methods, followed by delayed intervention with sclerotherapy. The primary outcomes will be frequency and severity of epistaxis. Secondary endpoints will be hemoglobin level, tolerability of treatment, additional treatment requirements, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of HHT based on the Curacoa Criteria
* age 18 and older
* cognitive ability and willingness to sign the study consent form and complete the study forms and questionnaires

Exclusion Criteria:

* previous sclerotherapy with Sodium Tetradecyl Sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Boyer, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Otolaryngology Clinic, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each group will get the same therapy in a different order Total number of subjects 18 with 2 incompletes. First period is 6 weeks with a 2 week washout period and 2 period is 6 weeks
Groups:
- Sclerotherapy Intervention Then Standard Treatment: This group will receive, on the first period of the study, sclerotherapy with STS to any visible lesions in the nose at the outset, followed by any needed standard treatments for breakthrough epistaxis. Washout period of 2 weeks
- Standard Treatment Then Sclerotherapy: The standard treatment group will continue their pre-study "standard treatment" methods to treat epistaxis on the first 6 weeks of the study, followed by intervention with sclerotherapy on the second 6 weeks of the study, plus any additionally needed standard treatments for breakthrough epistaxis. Wash out period 2 weeks
Period: Overall Study
Arm/Group | Sclerotherapy Intervention Then Standard Treatment | Standard Treatment Then Sclerotherapy
Started | 9 | 9
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 51.8 [31 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18
Curacao criteria [Number; unit: participants] — 1. Epistaxis;: spontaneous, recurrent nose bleeds 2. Telangiectases: multiple, at characteristic sites (lips, oral cavity, fingers, nose) 3. Visceral Lesions such as gastrointestinal telangiectasia (with or without bleeding), pulmonary arteriovenous malformation (AVM), hepatic AVM, cerebral AVMs, spinal AVM 4. Family history: a first degree relative with HHT according to these criteria
  Diagnosis of HHT Define: 3 criteria are present Possible or suspected: 2 criteria are present Unlikely: <2 criteria are present
  (Shovlin et al)
  participants
    Visceral Lesions | 9
    Family history: | 9
Number of Telangiectasia [Mean (Full Range); unit: Telangiectasia] | 7 [3 to 12]
Telangiectasia type [Number; unit: participants] — (I) isolated punctate telangiectasias or individual small arteriovenous malformation; (II) diffuse interconnecting vasculature with "feeder" vessels; and (III) large solitary arteriovenous malformation, which may be associated with scattered telangiectasia (Mahoney and Shapshay)
  participants
    Type 1 | 4
    Type 2 | 13
    Type 3 | 1
Prior Treatment [Number; unit: participants]
  Moisturization | 11
  Packing | 4
  Cautery | 3

OUTCOME MEASURES:

1. Primary Outcome: Severityof Epistaxis
Description: The primary outcome measure will be severity of epistaxis as measured by the Epistaxis Severity Score (ESS). The ESS, a recently developed online questionarrie that calculates the grading system for epistaxis severity. The higher the score the more severe the nose bleeds are Scale consists of several questions with a range of scale from 0-5 The average score is calculated for a final assessment
Time Frame: Change from Baseline to 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sclerotherapy Intervention: This group will receive, on the first period of the study, sclerotherapy with STS to any visible lesions in the nose at the outset, followed by any needed standard treatments for breakthrough epistaxis. On the second period of the study this group will continue with standard treatments that they had been receiving for epistaxis prior to the study. Standard treatment may include nasal packing, cauterization, laser treatments, microdebrider, and septodermoplasty.
  Sodium tetradecyl sulfate (sotradecol): 3% Sodium tetradecyl sulfate (STS) is mixed with air at a ratio of 4 parts air to 1 part STS for injection into the affected vessels in the nose. Topical anesthetic is applied to the nasal mucosa prior to injections. Once the mixture is ready for injection, the needle is placed into the vessel, in a submucosal fashion, penetrating 1-2 mm, and very small quantities of foam are injected
- Standard Treatment: The standard treatment group will continue their pre-study "standard treatment" methods to treat epistaxis on the first period of the study, followed by intervention with sclerotherapy on the second period of the study, plus any additionally needed standard treatments for breakthrough epistaxis. Standard treatment may include nasal packing, cauterization, laser treatments, microdebrider, septodermoplasty, and any other treatments that the patient reports using that are accepted as standard of care.
  Sodium tetradecyl sulfate (STS) is injected into the nasal lesions as a solution prepared by foaming STS with air at a 4:1 ratio. Individual injection amounts vary between lesions, patients and treatment sessions. No more than a total of 3 ml of solution is used in each session. Multiple lesions can be treated bilaterally, each with a separate injection.
  Standard Treatment
Arm/Group | Sclerotherapy Intervention | Standard Treatment
Number analyzed (Participants) | 16 | 16
units on a scale | -0.4578 (2.8943) | -1.4375 (4.1993)

ADVERSE EVENTS:
Groups:
- Sclerotherapy Intervention: This group will receive, on the first period of the study, sclerotherapy with STS to any visible lesions in the nose at the outset, followed by any needed standard treatments for breakthrough epistaxis. On the second period of the study this group will continue with standard treatments that they had been receiving for epistaxis prior to the study. Standard treatment may include nasal packing, cauterization, laser treatments, microdebrider, and septodermoplasty.
  Individual injection amounts vary between lesions, patients and treatment sessions. No more than 3 ml of solution is used in each session.
Arm/Group | Sclerotherapy Intervention | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No